CLINICAL TRIAL: NCT03385603
Title: The Role of Pain-related Fear in Sexual Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No individuals met eligibility or were enrolled.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201702214
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Sexual Pain Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive one of two treatments.
Who Masked: Investigator
Masking Description: An investigator who will not interact with study participants will perform the random intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fear-based Dilator Progression group (Experimental): Participants in this group will complete a home dilator program using levels of pain-related fear to progress through the program.
  Interventions: Device: Dilator; Behavioral: Fear-Based Questionnaires
- Standard Dilator Progression Group (Active Comparator): Participants in this group will complete a standard home program based on dilator manufacturer instructions for use.
  Interventions: Device: Dilator

INTERVENTIONS:
Device: Dilator — Both groups will have a home program consisting of dilators which are progressive in size. The standard care group will use manufacturer instructions to progress in size of dilators, while the experimental group will use self-reported levels of fear to progress in size of dilators.
Behavioral: Fear-Based Questionnaires — Series of questionnaires used to facilitate emotional awareness associated with vaginal and decreased sexual arousal.
  Arms: Fear-based Dilator Progression group

SUMMARY:
The purpose of this study is the evaluate the extent to which an intervention aimed at reducing pain-related fear affects sexual function and pain sensitivity compared to usual care.

DETAILED DESCRIPTION:
The overarching goal of this work is to identify the mechanisms underpinning sexual pain in women. Women with sexual pain exhibit higher vaginal pain sensitivity and lower levels of sexual desire and arousal compared to pain-free women. As a result of pain, sexual intercourse is avoided. Previous work in this area has examined a wide variety of interventions for sexual pain but has not examined how vaginal pain sensitivity and resulting sexual dysfunction may be mediated by pain-related fear. The study team proposes that a standardized exposure intervention that directly targets pain-related fear will in turn reduce vaginal pain sensitivity and translate to clinically meaningful changes in sexual function. The study team will assign women with sexual pain to receive a home-based, patient-controlled exposure intervention or standardized home-based home program. The specific aims of this proposal are: 1) To evaluate the extent to which pain-related fear mediates vaginal pain sensitivity in women with sexual pain; 2) To evaluate the extent to which graded exposure translates to changes in sexual function and partner dynamics. The completion of this work will provide us with a better understanding of the mechanisms underpinning sexual pain and specifically, how pain-related fear influences vaginal pain sensitivity and sexual function.

ELIGIBILITY:
Inclusion Criteria:

* Females with sexual pain >= 6 months
* Appropriate to use vaginal dilators
* The ability to read English and understand the informed consent form and screening questions
* The ability and willingness to follow all requirements of the study including following all directions and completion of daily pain reports
* Signed informed consent
* Are sexually active (have had intercourse at least twice in the last 30 days)
* Pain-related fear of intercourse greater than 50 on the numerical fear rating scale

Exclusion Criteria:

* Physical, psychological and medical issues, encountered during routine care that are felt insufficient for trial participation (physician discretion), such as poor mental status or neurological deficit limiting participation physically or cognitively (Mini-mental state exam less than 20).
* Women with sexual pain who are not sexually active (have not had intercourse at least twice in the last 30 days)
* Participants who use narcotic pain medication
* Participants diagnosed with a major depressive disorder
* Participants who exhibit signs and symptoms of infection, malignancy, or other conditions identified by a member of the study team that may be contraindications to the use of dilators
* Unable to readily access computer with Internet for reporting on daily fear levels and dilator size
* Pain-related fear of intercourse less than 50 on the numerical fear rating scale
* Women who are pregnant
* Participants who report a history of sexual abuse or trauma.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Vaginal Pain sensitivity | 40 days
  A change in pressure pain sensitivity at the vagina using a Wagner Digital Algometer.

SECONDARY OUTCOMES:
Sexual function | 40 days
  Assessed using the Female Sexual Function Index (FSFI), a 19- item questionnaire that measures desire, arousal, lubrication, orgasm, satisfaction, and pain in women with pelvic pain. This measure has high internal consistency (Cronbach's alpha 0.91-0.97) and good test-retest reliability (r=0.79-0.90).
Sexual Distress | 40 days
  Assessed using the Female Sexual Distress Scale-Revised (FSDS-R), a 13-item questionnaire that evaluates negative emotions about sexuality and sexual relations. The internal consistency of this measure is high (Cronbach's alpha 0.86- 0.94) with good test retest reliability (ICC= 0.74).
Partner dynamics | 40 days
  Assessed using the Revised Dyadic Adjustment Scale(RDAS), a 14-item questionnaire that assesses three overarching dimensions of relationships, including Consensus, Satisfaction, and Cohesion. This measure has high internal consistency (Cronbach's alpha= 0.90).

CONTACTS AND LOCATIONS:
Overall Officials: Meryl Alappattu, DPT, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health at Springhill, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No